CLINICAL TRIAL: NCT02201524
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study To Evaluate Safety And Efficacy Of Pf-04965842 In Subjects With Moderate To Severe Psoriasis
Brief Title: Study to Evaluate PF-04965842 in Patients With Moderate to Severe Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated 26 June 2015 due to changes in the drug development portfolio. This study was not terminated for reasons of safety and/or efficacy
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7451005; JAK-1 FOR PSORIASIS (Other: Alias Study Number)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Plaque Psoriasis
Keywords: Phase 2; randomized; double-blind; placebo; plaque; psoriasis; safety; efficacy; JAK; janus kinase; moderate; severe
MeSH Terms: conditions — Plaque, Amyloid; Psoriasis; Lymphoma, Follicular | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 200mg of PF-04965842 twice daily
  Interventions: Drug: PF-04965842
- Cohort 2 (Experimental): 400mg of PF-04965842 once daily
  Interventions: Drug: PF-04965842
- Cohort 3 (Experimental): 200mg of PF-04965842 once daily
  Interventions: Drug: PF-04965842
- Cohort 4 (Placebo Comparator): Placebo comparator daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-04965842 — Subjects will receive 200 mg PF 04965842 twice daily for 4 weeks
  Other Names: JAK1 inhibitor
  Arms: Cohort 1
Drug: PF-04965842 — Subjects will receive 400 mg PF 04965842 daily for 4 weeks
  Other Names: JAK1 inhibitor
  Arms: Cohort 2
Drug: PF-04965842 — Subjects will receive 200 mg PF 04965842 daily for 4 weeks
  Other Names: JAK1 inhibitor
  Arms: Cohort 3
Other: Placebo — Subjects will receive placebo for 4 weeks
  Arms: Cohort 4

SUMMARY:
Study B7451005 is a Phase 2 study which will assess the efficacy and safety of PF-04965842 in patients with moderate to severe psoriasis. The study will include three PF-04965842 groups (200 mg daily, 400 mg daily and 200 mg twice daily) and a placebo group. The treatment period will be 4 weeks in duration and will be followed up by a 4 week follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of plaque psoriasis for at least 6 months prior to first study dose.
2. Have plaque type psoriasis covering at least 15% of total BSA at Day 1 (at the time of the first study dose).
3. Have a PASI score of 12 or greater at Day 1 (at the time of the first study dose).
4. Be a candidate for phototherapy or systemic treatment of psoriasis (either naïve or history of previous treatment).

Exclusion Criteria:

1. Currently have non plaque forms of psoriasis, eg, erythrodermic, guttate, or pustular psoriasis.
2. 3. Have current drug induced psoriasis, eg, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, antimalarial drugs or lithium.
3. Have received any of the following treatment regimens specified in the timeframes outlined below:

Within 9 months of first dose of study drug:

• Ustekinumab (Stelara).

Within 12 weeks of first dose of study drug:

• Any experimental therapy for psoriasis or rheumatoid arthritis.

Within 4 8 weeks of first dose of study drug:

* Biologic therapies for psoriasis have discontinuation periods determined from approximately 5x half life of the respective biologic:
* 4 weeks: etanercept (Enbrel).
* 8 weeks: infliximab (Remicade), adalimumab (Humira).

Within 4 weeks of first dose of study drug:

* Systemic treatments other than biologics that could affect psoriasis (eg, oral or injectable corticosteroids, retinoids, methotrexate, cyclosporine, fumaric acid derivatives, sulfasalazine, hydroxycarbamide (hydroxyurea), azathioprine).
* Phototherapy and psoralen plus ultraviolet A therapy (PUVA).
* Other - intramuscular gold, immunization with any live virus vaccination (eg, FluMist), herbal medications.

Within 2 weeks of first dose of study drug:

* Topical treatments that could affect psoriasis (eg, corticosteroids, tars, keratolytics, anthralin, vitamin D analogs, and retinoids).
* Phototherapy with ultraviolet B (UVB) (narrowband or broadband).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (35):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Northwest Arkansas Clinical Trials Center, PLLC/Hull Dermatology, PA, Rogers, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Huntington Medical Foundation/Specialty Office, Pasadena, California
  - Clinical Science Institute, Santa Monica, California
  - Olympian Clinical Research, Clearwater, Florida
  - Westcoast Radiology Services, Clearwater, Florida
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Ormond Beach, Florida
  - Advanced Medical Research, Inc, Atlanta, Georgia
  - Columbus Dermatology, P.C., Columbus, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - DS Research, Louisville, Kentucky
  - Shondra L Smith, MD, Lake Charles, Louisiana
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center - Section of Dermatology, Lebanon, New Hampshire
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center - Shipment Only, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Health Concepts, Rapid City, South Dakota
  - Arlington Research Center, Inc., Arlington, Texas
  - Dermatology Treatment & Research Center, PA, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Virginia Clinical Research, Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington
- Canada (10):
  - Enverus Medical Research, Surrey, British Columbia
  - Co-Medica Research Network Inc., Courtice, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Research by ICLS, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology & Cosmetic, Richmond Hill, Ontario
  - K.Papp Clinical Research Inc., Waterloo, Ontario
  - Dr Isabelle Delorme Inc., Drummondville, Quebec
  - Innovaderm Research Inc., Montreal, Quebec
  - Q & T Research Sherbrooke Inc., Sherbrooke, Quebec

REFERENCES:
- [Derived] Armstrong AW, Alexis AF, Blauvelt A, Silverberg JI, Feeney C, Levenberg M, Chan G, Zhang F, Fostvedt L. Predicting Abrocitinib Efficacy at Week 12 Based on Clinical Response at Week 4: A Post Hoc Analysis of Four Randomized Studies in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1849-1861. doi: 10.1007/s13555-024-01183-3. Epub 2024 Jun 19. PMID 38896380
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population pharmacokinetic-pharmacodynamic modelling of platelet time-courses following administration of abrocitinib. Br J Clin Pharmacol. 2022 Aug;88(8):3856-3871. doi: 10.1111/bcp.15334. Epub 2022 Apr 11. PMID 35342978
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7451005&StudyName=Study%20to%20evaluate%20PF-04965842%20in%20Patients%20with%20Moderate%20to%20Severe%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to PF-04965842 tablets orally from Day 1 to 28.
- PF-04965842 200 Milligram (mg) Once Daily: Participants received PF-04965842 200 mg tablets, orally once daily from Day 1 to 28.
- PF-04965842 400 mg Once Daily: Participants received PF-04965842 400 mg tablets, orally once daily from Days 1 to 28.
- PF-04965842 200 mg Twice Daily: Participants received PF-04965842 200 mg tablets, orally twice daily from Day 1 to 28.
Period: Overall Study
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Started | 14 | 15 | 16 | 14
Completed | 12 | 12 | 12 | 10
Not Completed | 2 | 3 | 4 | 4
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Insufficient clinical response | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — No longer meets eligibility criteria | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Other | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of the randomized study drug (PF-04965842 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily | Total
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (10.8) | 42.9 (12.3) | 42.8 (11.6) | 52.1 (9.7) | 45.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 6 | 19
  Male | 11 | 10 | 11 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 4
Description: PASI score is the combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated: 0 (no involvement) to 6 (90-100 percent involvement), severity estimated by clinical signs: erythema (E), induration (I), scaling (S); 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4).
Time Frame: Baseline, Week 4
Population: The modified intent to treat (mITT) analysis set included all randomized participants who received at least 1 dose of the randomized study drug (PF-04965842 or placebo). Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
units on a scale
  Baseline (n= 14, 15, 16, 14) | 20.05 (3.993) | 20.34 (7.089) | 19.21 (4.426) | 18.01 (5.507)
  Change at Week 4 (n= 12, 12, 12, 10) | -6.61 (7.252) | -11.73 (6.658) | -13.09 (7.979) | -13.71 (6.248)
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo: Longitudinal analysis of covariance (LANCOVA) model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; Least square (LS) mean difference = -5.08, 90% CI 2-sided [-9.15 to -1.01], Standard Error of Mean 2.420
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -5.61, 90% CI 2-sided [-9.61 to -1.62], Standard Error of Mean 2.375
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -9.98, 90% CI 2-sided [-14.19 to -5.77], Standard Error of Mean 2.506

2. Secondary Outcome: Percent Change From Baseline in PASI Score at Week 1, 2, 3, 4, 5, 6, and 8
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 8
Population: The mITT analysis set included all randomized participants who received at least 1 dose of the randomized study drug. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
percent change
  Change at Week 1 (n= 14, 15, 16, 14) | -13.68 (18.527) | -23.27 (18.796) | -24.07 (22.272) | -30.99 (28.557)
  Change at Week 2 (n= 14, 14, 13, 12) | -26.68 (25.776) | -27.96 (20.161) | -41.54 (28.779) | -49.09 (30.153)
  Change at Week 3 (n= 13, 12, 15, 11) | -27.06 (31.220) | -33.96 (19.793) | -53.18 (33.326) | -73.37 (22.569)
  Change at Week 4 (n= 12, 12, 12, 10) | -33.59 (31.574) | -57.61 (21.594) | -64.46 (32.175) | -80.96 (23.155)
  Change at Week 5 (n= 11, 12, 12, 9) | -42.62 (21.228) | -58.63 (16.015) | -57.76 (37.397) | -80.80 (20.279)
  Change at Week 6 (n= 11, 11, 10, 10) | -39.85 (28.661) | -61.02 (11.655) | -56.94 (39.558) | -69.15 (26.871)
  Change at Week 8 (n= 8, 11, 11, 8) | -44.62 (26.616) | -44.28 (27.486) | -48.63 (35.373) | -61.67 (29.352)
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 1: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -9.32, 90% CI 2-sided [-23.19 to 4.56], Standard Error of Mean 8.291
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 1: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -11.19, 90% CI 2-sided [-24.87 to 2.50], Standard Error of Mean 8.177
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -19.22, 90% CI 2-sided [-33.45 to -4.99], Standard Error of Mean 8.504
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 2: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -4.30, 90% CI 2-sided [-21.71 to 13.11], Standard Error of Mean 10.387
Statistical Analysis 5: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 2: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -18.04, 90% CI 2-sided [-35.25 to -0.82], Standard Error of Mean 10.273
Statistical Analysis 6: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -27.07, 90% CI 2-sided [-44.90 to -9.23], Standard Error of Mean 10.646
Statistical Analysis 7: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 3: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -10.07, 90% CI 2-sided [-28.53 to 8.39], Standard Error of Mean 11.013
Statistical Analysis 8: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 3: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -29.23, 90% CI 2-sided [-47.33 to -11.13], Standard Error of Mean 10.793
Statistical Analysis 9: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; LS mean difference = -49.99, 90% CI 2-sided [-68.92 to -31.05], Standard Error of Mean 11.299
Statistical Analysis 10: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 4: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -24.25, 90% CI 2-sided [-43.26 to -5.24], Standard Error of Mean 11.330
Statistical Analysis 11: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 4: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -27.47, 90% CI 2-sided [-46.18 to -8.75], Standard Error of Mean 11.155
Statistical Analysis 12: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; LS mean difference = -52.63, 90% CI 2-sided [-72.24 to -33.02], Standard Error of Mean 11.697
Statistical Analysis 13: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 5: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LANCOVA; LS mean difference = -17.98, 90% CI 2-sided [-35.80 to -0.15], Standard Error of Mean 10.605
Statistical Analysis 14: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 5: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -14.78, 90% CI 2-sided [-32.44 to 2.88], Standard Error of Mean 10.513
Statistical Analysis 15: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; LS mean difference = -47.94, 90% CI 2-sided [-66.61 to -29.27], Standard Error of Mean 11.125
Statistical Analysis 16: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 6: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean = -21.75, 90% CI 2-sided [-41.00 to -2.49], Standard Error of Mean 11.459
Statistical Analysis 17: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 6: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -17.75, 90% CI 2-sided [-36.92 to 1.42], Standard Error of Mean 11.416
Statistical Analysis 18: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; LS mean difference = -35.88, 90% CI 2-sided [-55.85 to -15.90], Standard Error of Mean 11.893
Statistical Analysis 19: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 8: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -10.75, 90% CI 2-sided [-32.57 to 11.07], Standard Error of Mean 12.985
Statistical Analysis 20: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 8: LANCOVA model contains fixed factors of treatment, week, treatment by week interaction, baseline value and unstructured covariance matrix; Test type: Superiority or Other; LS mean difference = -13.03, 90% CI 2-sided [-34.71 to 8.64], Standard Error of Mean 12.902
Statistical Analysis 21: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; LS mean difference = -34.46, 90% CI 2-sided [-57.44 to -11.48], Standard Error of Mean 13.690

3. Secondary Outcome: Change From Baseline in PASI Score at Week 1, 2, 3, 5, 6 and 8
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2, 3, 5, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
units on a scale
  Change at Week 1 (n= 14, 15, 16, 14) | -2.96 (4.306) | -5.13 (4.902) | -4.79 (4.900) | -5.46 (4.965)
  Change at Week 2 (n= 14, 14, 13, 12) | -5.26 (5.205) | -5.80 (4.915) | -8.33 (7.103) | -8.51 (5.860)
  Change at Week 3 (n= 13, 12, 15, 11) | -5.38 (7.033) | -7.44 (5.824) | -10.77 (8.048) | -12.61 (4.461)
  Change at Week 5 (n= 11, 12, 12, 9) | -8.69 (5.314) | -11.68 (5.262) | -11.77 (8.421) | -14.17 (6.483)
  Change at Week 6 (n= 11, 11, 10, 10) | -8.05 (6.989) | -12.00 (4.901) | -12.13 (9.576) | -11.80 (6.678)
  Change at Week 8 (n= 8, 11, 11, 8) | -9.33 (6.745) | -8.38 (4.933) | -10.04 (8.287) | -10.75 (6.382)
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -2.01, 90% CI 2-sided [-4.73 to 0.72], Standard Error of Mean 1.626
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 400 mg Once Daily; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -2.31, 90% CI 2-sided [-4.99 to 0.38], Standard Error of Mean 1.603
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -3.65, 90% CI 2-sided [-6.45 to -0.86], Standard Error of Mean 1.668
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -1.08, 90% CI 2-sided [-4.49 to 2.32], Standard Error of Mean 2.032
Statistical Analysis 5: Comparison: Placebo vs PF-04965842 400 mg Once Daily; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; LS mean difference = -3.86, 90% CI 2-sided [-7.23 to -0.49], Standard Error of Mean 2.011
Statistical Analysis 6: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -5.16, 90% CI 2-sided [-8.65 to -1.67], Standard Error of Mean 2.084
Statistical Analysis 7: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; LS mean difference = -2.34, 90% CI 2-sided [-6.07 to 1.39], Standard Error of Mean 2.224
Statistical Analysis 8: Comparison: Placebo vs PF-04965842 400 mg Once Daily; [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; LS mean difference = -6.12, 90% CI 2-sided [-9.78 to -2.47], Standard Error of Mean 2.177
Statistical Analysis 9: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; LS mean difference = -9.39, 90% CI 2-sided [-13.22 to -5.56], Standard Error of Mean 2.286
Statistical Analysis 10: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; LS mean difference = -3.25, 90% CI 2-sided [-6.71 to 0.21], Standard Error of Mean 2.054
Statistical Analysis 11: Comparison: Placebo vs PF-04965842 400 mg Once Daily; [analysis description as in outcome 2, analysis 14]; Test type: Superiority or Other; LS mean difference = -2.98, 90% CI 2-sided [-6.40 to 0.45], Standard Error of Mean 2.035
Statistical Analysis 12: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; LS mean difference = -8.59, 90% CI 2-sided [-12.24 to -4.95], Standard Error of Mean 2.167
Statistical Analysis 13: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; LS mean difference = -3.98, 90% CI 2-sided [-7.89 to -0.08], Standard Error of Mean 2.321
Statistical Analysis 14: Comparison: Placebo vs PF-04965842 400 mg Once Daily; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; LS mean difference = -3.80, 90% CI 2-sided [-7.68 to 0.07], Standard Error of Mean 2.304
Statistical Analysis 15: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; LS mean difference = -6.94, 90% CI 2-sided [-11.00 to -2.89], Standard Error of Mean 2.412
Statistical Analysis 16: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; LS mean difference = -1.27, 90% CI 2-sided [-5.65 to 3.11], Standard Error of Mean 2.607
Statistical Analysis 17: Comparison: Placebo vs PF-04965842 400 mg Once Daily; [analysis description as in outcome 2, analysis 20]; Test type: Superiority or Other; LS mean difference = -2.83, 90% CI 2-sided [-7.18 to 1.51], Standard Error of Mean 2.586
Statistical Analysis 18: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; LS mean difference = -6.52, 90% CI 2-sided [-11.15 to -1.89], Standard Error of Mean 2.758

4. Secondary Outcome: Percentage of Participants Achieving 50 Percent Reduction From Baseline PASI Score at Week 1, 2, 3, 4, 5, 6, and 8
Description: PASI score is combined assessment of lesion severity and area affected into single score range:0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated:0 (no involvement) to 6 (90-100 percent involvement), severity estimated by clinical signs: erythema (E), induration (I), scaling (S); 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4). Participants who had at least 50 percent reduction in PASI score relative to baseline PASI Score are reported. 90 percent confidence intervals are calculated using clopper-pearson (exact) method.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 8
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
percentage of participants
  Week 1 (n= 14, 15, 16, 14) | 7.1 [0.4 to 29.7] | 6.7 [0.3 to 27.9] | 25.0 [9.0 to 48.4] | 21.4 [6.1 to 46.6]
  Week 2 (n= 14, 14, 13, 12) | 21.4 [6.1 to 46.6] | 7.1 [0.4 to 29.7] | 23.1 [6.6 to 49.5] | 41.7 [18.1 to 68.5]
  Week 3 (n= 13, 12, 15, 11) | 23.1 [6.6 to 49.5] | 25.0 [7.2 to 52.7] | 46.7 [24.4 to 70.0] | 90.9 [63.6 to 99.5]
  Week 4 (n= 12, 12, 12, 10) | 25.0 [7.2 to 52.7] | 66.7 [39.1 to 87.7] | 66.7 [39.1 to 87.7] | 80.0 [49.3 to 96.3]
  Week 5 (n= 11, 12, 12, 9) | 54.5 [27.1 to 80.0] | 66.7 [39.1 to 87.7] | 58.3 [31.5 to 81.9] | 100.0 [71.7 to 100]
  Week 6 (n= 11, 11, 10, 10) | 45.5 [20.0 to 72.9] | 81.8 [53.0 to 96.7] | 60.0 [30.4 to 85.0] | 70.0 [39.3 to 91.3]
  Week 8 (n= 8, 11, 11, 8) | 50.0 [19.3 to 80.7] | 45.5 [20.0 to 72.9] | 63.6 [35.0 to 86.5] | 62.5 [28.9 to 88.9]
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 1: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -0.5, 90% CI 2-sided [-21.5 to 19.6]
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 1: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 17.9, 90% CI 2-sided [-5.9 to 40.3]
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 1: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage Analysed using; Difference in Percentage = 14.3, 90% CI 2-sided [-9.3 to 38.0]
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -14.3, 90% CI 2-sided [-38.0 to 9.3]
Statistical Analysis 5: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 1.6, 90% CI 2-sided [-25.4 to 29.1]
Statistical Analysis 6: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 20.2, 90% CI 2-sided [-10.2 to 48.3]
Statistical Analysis 7: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 1.9, 90% CI 2-sided [-26.7 to 31.0]
Statistical Analysis 8: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 23.6, 90% CI 2-sided [-6.9 to 49.8]
Statistical Analysis 9: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 67.8, 90% CI 2-sided [36.4 to 85.3]
Statistical Analysis 10: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 41.7, 90% CI 2-sided [7.6 to 67.1]
Statistical Analysis 11: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 41.7, 90% CI 2-sided [7.6 to 67.1]
Statistical Analysis 12: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 55.0, 90% CI 2-sided [19.7 to 77.6]
Statistical Analysis 13: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 12.1, 90% CI 2-sided [-21.4 to 43.4]
Statistical Analysis 14: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 3.8, 90% CI 2-sided [-29.4 to 36.4]
Statistical Analysis 15: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 45.5, 90% CI 2-sided [17.1 to 69.0]
Statistical Analysis 16: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 36.4, 90% CI 2-sided [1.9 to 63.4]
Statistical Analysis 17: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 14.5, 90% CI 2-sided [-21.4 to 47.0]
Statistical Analysis 18: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 24.5, 90% CI 2-sided [-11.8 to 54.9]
Statistical Analysis 19: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -4.5, 90% CI 2-sided [-40.4 to 32.3]
Statistical Analysis 20: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 13.6, 90% CI 2-sided [-23.7 to 48.2]
Statistical Analysis 21: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 12.5, 90% CI 2-sided [-28.0 to 49.3]

5. Secondary Outcome: Percentage of Participants Achieving 75 Percent Reduction From Baseline PASI Score at Week 1, 2, 3, 4, 5, 6 and 8
Description: PASI score is combined assessment of lesion severity and area affected into single score range:0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated:0 (no involvement) to 6 (90-100 percent involvement), severity estimated by clinical signs: erythema (E), induration (I), scaling (S); 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4). Participants who had at least 75 percent reduction in PASI score relative to baseline PASI Score are reported. 90 percent confidence intervals are calculated using clopper-pearson (exact) method.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 8
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
percentage of participants
  Week 1 (n= 14, 15, 16, 14) | 0.0 [0.0 to 19.3] | 0.0 [0.0 to 18.1] | 0.0 [0.0 to 17.1] | 7.1 [0.4 to 29.7]
  Week 2 (n= 14, 14, 13, 12) | 7.1 [0.4 to 29.7] | 0.0 [0.0 to 19.3] | 15.4 [2.8 to 41.0] | 25.0 [7.2 to 52.7]
  Week 3 (n= 13, 12, 15, 11) | 7.7 [0.4 to 31.6] | 0.0 [0.0 to 22.1] | 40.0 [19.1 to 64.0] | 36.4 [13.5 to 65.0]
  Week 4 (n= 12, 12, 12, 10) | 16.7 [3.0 to 43.8] | 16.7 [3.0 to 43.8] | 50.0 [24.5 to 75.5] | 60.0 [30.4 to 85.0]
  Week 5 (n= 11, 12, 12, 9) | 0.0 [0.0 to 23.8] | 25.0 [7.2 to 52.7] | 50.0 [24.5 to 75.5] | 66.7 [34.5 to 90.2]
  Week 6 (n= 11, 11, 10, 10) | 18.2 [3.3 to 47.0] | 9.1 [0.5 to 36.4] | 60.0 [30.4 to 85.0] | 50.0 [22.2 to 77.8]
  Week 8 (n= 8, 11, 11, 8) | 25.0 [4.6 to 60.0] | 9.1 [0.5 to 36.4] | 18.2 [3.3 to 47.0] | 25.0 [4.6 to 60.0]
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 1: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 7.1, 90% CI 2-sided [-10.2 to 27.0]
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -7.1, 90% CI 2-sided [-27.0 to 10.2]
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 8.2, 90% CI 2-sided [-14.4 to 32.2]
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 17.9, 90% CI 2-sided [-6.7 to 43.6]
Statistical Analysis 5: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -7.7, 90% CI 2-sided [-28.8 to 12.1]
Statistical Analysis 6: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 32.3, 90% CI 2-sided [5.4 to 55.4]
Statistical Analysis 7: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 28.7, 90% CI 2-sided [0.8 to 55.3]
Statistical Analysis 8: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 0.0, 90% CI 2-sided [-27.3 to 27.3]
Statistical Analysis 9: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 33.3, 90% CI 2-sided [1.0 to 59.8]
Statistical Analysis 10: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 43.3, 90% CI 2-sided [8.8 to 69.3]
Statistical Analysis 11: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 25.0, 90% CI 2-sided [2.1 to 49.3]
Statistical Analysis 12: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 50.0, 90% CI 2-sided [25.4 to 71.8]
Statistical Analysis 13: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 66.7, 90% CI 2-sided [39.2 to 86.1]
Statistical Analysis 14: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -9.1, 90% CI 2-sided [-36.3 to 18.3]
Statistical Analysis 15: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 41.8, 90% CI 2-sided [6.2 to 68.5]
Statistical Analysis 16: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 31.8, 90% CI 2-sided [-2.9 to 60.5]
Statistical Analysis 17: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -15.9, 90% CI 2-sided [-47.8 to 13.7]
Statistical Analysis 18: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -6.8, 90% CI 2-sided [-40.6 to 24.8]
Statistical Analysis 19: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 0.0, 90% CI 2-sided [-36.4 to 36.4]

6. Secondary Outcome: Percentage of Participants Achieving 90 Percent Reduction From Baseline PASI Score at Week 1, 2, 3, 4, 5, 6, and 8
Description: PASI score is combined assessment of lesion severity and area affected into single score range:0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated:0 (no involvement) to 6 (90-100 percent involvement), severity estimated by clinical signs: erythema (E), induration (I), scaling (S); 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4). Participants who had at least 90 percent reduction in PASI score relative to baseline PASI Score are reported. 90 percent confidence intervals are calculated using clopper-pearson (exact) method.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 8 (early termination)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
percentage of participants
  Week 1 (n= 14, 15, 16, 14) | 0.0 [0.0 to 19.3] | 0.0 [0.0 to 18.1] | 0.0 [0.0 to 17.1] | 7.1 [0.4 to 29.7]
  Week 2 (n= 14, 14, 13, 12) | 7.1 [0.4 to 29.7] | 0.0 [0.0 to 19.3] | 7.7 [0.4 to 31.6] | 8.3 [0.4 to 33.9]
  Week 3 (n= 13, 12, 15, 11) | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 22.1] | 13.3 [2.4 to 36.3] | 36.4 [13.5 to 65.0]
  Week 4 (n= 12, 12, 12, 10) | 0.0 [0.0 to 22.1] | 0.0 [0.0 to 22.1] | 33.3 [12.3 to 60.9] | 60.0 [30.4 to 85.0]
  Week 5 (n= 11, 12, 12, 9) | 0.0 [0.0 to 23.8] | 0.0 [0.0 to 22.1] | 25.0 [7.2 to 52.7] | 44.4 [16.9 to 74.9]
  Week 6 (n= 11, 11, 10, 10) | 0.0 [0.0 to 23.8] | 0.0 [0.0 to 23.8] | 20.0 [3.7 to 50.7] | 30.0 [8.7 to 60.7]
  Week 8 (n= 8, 11, 11, 8) | 0.0 [0.0 to 31.2] | 0.0 [0.0 to 23.8] | 0.0 [0.0 to 23.8] | 25.0 [4.6 to 60.0]
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 1: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 7.1, 90% CI 2-sided [-10.2 to 27.0]
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = -7.1, 90% CI 2-sided [-27.0 to 10.2]
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 0.5, 90% CI 2-sided [-20.7 to 22.8]
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 1.2, 90% CI 2-sided [-20.3 to 24.8]
Statistical Analysis 5: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 13.3, 90% CI 2-sided [-5.6 to 33.8]
Statistical Analysis 6: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 36.4, 90% CI 2-sided [15.3 to 61.1]
Statistical Analysis 7: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 33.3, 90% CI 2-sided [11.3 to 57.3]
Statistical Analysis 8: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 60.0, 90% CI 2-sided [34.7 to 80.9]
Statistical Analysis 9: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 25.0, 90% CI 2-sided [2.1 to 49.3]
Statistical Analysis 10: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 44.4, 90% CI 2-sided [19.4 to 70.2]
Statistical Analysis 11: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 20.0, 90% CI 2-sided [-2.7 to 46.6]
Statistical Analysis 12: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 30.0, 90% CI 2-sided [6.4 to 56.4]
Statistical Analysis 13: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 25.0, 90% CI 2-sided [-4.9 to 54.9]

7. Secondary Outcome: Percentage of Participants Achieving Physician Global Assessment (PGA) Response of 'Clear' or 'Almost Clear' at Week 1, 2, 3, 4, 5, 6, and 8
Description: The PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema (E), induration (I), and scaling (S) across all psoriatic lesions. The severity rating scores (erythema: 0= no evidence of erythema to 4= dark, deep red; Induration: 0= no evidence of plaque elevation to 4= marked plaque elevation, hard/sharp borders; Scaling: 0= no evidence of scaling to 4= thick, coarse scale predominates) were summed (E + I + S= total) and the average (total/3) was taken. The total average was rounded to the nearest whole number score to determine the PGA. The 5-point scale for PGA was: 0= clear; 1= almost clear; 2= mild; 3= moderate; 4= severe, where higher score indicating more severity. Participants with response of clear and almost clear were reported. 90 percent confidence intervals were calculated using clopper-pearson (exact) method.
Time Frame: Week 1, 2, 3, 4, 5, 6, 8
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
percentage of participants
  Week 1 (n= 14, 15, 16, 14) | 0.0 [0.0 to 19.3] | 13.3 [2.4 to 36.3] | 12.5 [2.3 to 34.4] | 7.1 [0.4 to 29.7]
  Week 2 (n= 14, 14, 13, 12) | 7.1 [0.4 to 29.7] | 28.6 [10.4 to 54.0] | 23.1 [6.6 to 49.5] | 41.7 [18.1 to 68.5]
  Week 3 (n= 13, 12, 15, 11) | 15.4 [2.8 to 41.0] | 33.3 [12.3 to 60.9] | 46.7 [24.4 to 70.0] | 45.5 [20.0 to 72.9]
  Week 4 (n= 12, 12, 12, 10) | 16.7 [3.0 to 43.8] | 41.7 [18.1 to 68.5] | 58.3 [31.5 to 81.9] | 70.0 [39.3 to 91.3]
  Week 5 (n= 11, 12, 12, 9) | 27.3 [7.9 to 56.4] | 33.3 [12.3 to 60.9] | 41.7 [18.1 to 68.5] | 77.8 [45.0 to 95.9]
  Week 6 (n= 11, 11, 10, 10) | 36.4 [13.5 to 65.0] | 45.5 [20.0 to 72.9] | 40.0 [15.0 to 69.6] | 50.0 [22.2 to 77.8]
  Week 8 (n= 8, 11, 11, 8) | 25.0 [4.6 to 60.0] | 27.3 [7.9 to 56.4] | 45.5 [20.0 to 72.9] | 37.5 [11.1 to 71.1]
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 1: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 13.3, 90% CI 2-sided [-4.4 to 33.8]
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 1: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 12.5, 90% CI 2-sided [-5.2 to 32.0]
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 1: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 7.1, 90% CI 2-sided [-10.2 to 27.0]
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 21.4, 90% CI 2-sided [-3.2 to 45.5]
Statistical Analysis 5: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 15.9, 90% CI 2-sided [-8.1 to 40.7]
Statistical Analysis 6: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 2: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 34.5, 90% CI 2-sided [7.3 to 59.4]
Statistical Analysis 7: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 17.9, 90% CI 2-sided [-11.2 to 45.5]
Statistical Analysis 8: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 31.3, 90% CI 2-sided [1.7 to 55.7]
Statistical Analysis 9: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 3: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage Analysed using; Difference in Percentage = 30.1, 90% CI 2-sided [-1.2 to 57.4]
Statistical Analysis 10: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 25.0, 90% CI 2-sided [-6.4 to 52.5]
Statistical Analysis 11: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 41.7, 90% CI 2-sided [8.7 to 66.7]
Statistical Analysis 12: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 4: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 53.3, 90% CI 2-sided [18.5 to 76.6]
Statistical Analysis 13: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 6.1, 90% CI 2-sided [-26.1 to 36.6]
Statistical Analysis 14: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 14.4, 90% CI 2-sided [-18.9 to 44.5]
Statistical Analysis 15: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 5: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 50.5, 90% CI 2-sided [12.9 to 75.3]
Statistical Analysis 16: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 9.1, 90% CI 2-sided [-25.2 to 41.4]
Statistical Analysis 17: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 3.6, 90% CI 2-sided [-30.5 to 37.3]
Statistical Analysis 18: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 6: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 13.6, 90% CI 2-sided [-21.9 to 46.2]
Statistical Analysis 19: Comparison: Placebo vs PF-04965842 200 Milligram (mg) Once Daily; PF-04965842 200 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 2.3, 90% CI 2-sided [-33.2 to 34.6]
Statistical Analysis 20: Comparison: Placebo vs PF-04965842 400 mg Once Daily; PF-04965842 400 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 20.5, 90% CI 2-sided [-17.6 to 51.9]
Statistical Analysis 21: Comparison: Placebo vs PF-04965842 200 mg Twice Daily; PF-04965842 200 mg vs Placebo at Week 8: Analysed using Asymptotic Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentage = 12.5, 90% CI 2-sided [-26.4 to 48.1]

8. Secondary Outcome: Change From Baseline in Fasting Lipids at Week 2, 4 and 8
Description: Participants were required to fast 9 hours prior to sampling for lipid profile which included following parameters: low-density lipoprotein-cholesterol (LDL-C), high-density lipoprotein-cholesterol (HDL-C), cholesterol, triglycerides.
Time Frame: Baseline, Week 2, 4, 8 (early termination)
Population: The safety analysis population set included all enrolled participants who received at least 1 dose of study drug. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
milligram per deciliter (mg/dL)
  Baseline: (n= 14, 15. 16, 14) | 119.07 (24.780) [107.34 to 130.80] | 105.27 (28.632) [92.25 to 118.29] | 114.56 (28.317) [102.15 to 126.97] | 113.93 (31.770) [98.89 to 128.97]
  LDL-C: Change at Week 2 (n= 13, 14, 14, 12) | -6.31 (16.825) [-14.62 to 2.01] | 18.50 (31.035) [3.81 to 33.19] | 3.21 (25.097) [-8.66 to 15.09] | 26.92 (24.748) [14.09 to 39.75]
  LDL-C: Change at Week 4 (n= 12, 12, 12, 10) | -2.50 (11.350) [-8.38 to 3.38] | 26.75 (26.455) [13.04 to 40.46] | 10.17 (22.143) [-1.31 to 21.65] | 15.20 (30.904) [-2.71 to 33.11]
  LDL-C: Change at Week 8 (n= 7, 11, 10, 8) | 7.14 (20.659) [-8.03 to 22.32] | 6.00 (16.529) [-3.03 to 15.03] | -3.20 (12.072) [-10.20 to 3.80] | -15.13 (20.301) [-28.72 to -1.53]
  HDL-C: Baseline (n= 14, 15, 16, 14) | 52.93 (12.640) [46.95 to 58.91] | 46.47 (11.230) [41.36 to 51.57] | 49.06 (15.058) [42.46 to 55.66] | 50.29 (10.163) [45.48 to 55.10]
  HDL-C: Change at Week 2 (n= 13, 14, 14, 12) | -1.54 (7.881) [-5.43 to 2.36] | 10.00 (5.533) [7.38 to 12.62] | 10.64 (9.295) [6.24 to 15.04] | 14.00 (8.113) [9.79 to 18.21]
  HDL-C: Change at Week 4 (n= 12, 12, 12, 10) | -1.00 (6.238) [-4.23 to 2.23] | 9.25 (6.717) [5.77 to 12.73] | 12.25 (10.437) [6.84 to 17.66] | 12.80 (10.075) [6.96 to 18.64]
  HDL-C: Change at Week 8 (n= 7, 11, 10, 8) | -2.43 (10.737) [-10.31 to 5.46] | -2.36 (2.730) [-3.86 to -0.87] | -0.40 (6.275) [-4.04 to 3.24] | -5.00 (6.234) [-9.18 to -0.82]
  Cholesterol: Baseline (n= 14, 15, 16, 14) | 195.43 (30.137) [181.16 to 209.69] | 186.80 (25.741) [175.09 to 198.51] | 188.75 (32.298) [174.60 to 202.90] | 191.14 (36.469) [173.88 to 208.40]
  Cholesterol: Change at Week 2 (n= 13, 14, 14 12) | -0.77 (14.800) [-8.08 to 6.55] | 29.57 (31.329) [14.74 to 44.40] | 21.00 (34.005) [4.91 to 37.09] | 44.08 (23.469) [31.92 to 56.25]
  Cholesterol: Change at Week 4 (n= 12, 12, 12, 10) | -3.50 (20.174) [-13.96 to 6.96] | 40.08 (25.062) [27.09 to 53.08] | 27.25 (22.919) [15.37 to 39.13] | 26.40 (29.220) [9.46 to 43.34]
  Cholesterol: Change at Week 8 (n= 7, 11, 10, 8) | 9.86 (24.361) [-8.04 to 27.75] | 7.45 (14.733) [-0.60 to 15.51] | -1.20 (20.395) [-13.02 to 10.62] | -10.88 (23.991) [-26.94 to 5.19]
  Triglycerides: Baseline (n= 14, 15, 16, 14) | 116.64 (47.490) [94.17 to 139.12] | 175.00 (74.971) [140.91 to 209.09] | 125.50 (50.552) [103.35 to 147.65] | 134.21 (53.903) [108.70 to 159.73]
  Triglycerides: Change at Week 2 (n= 13, 14, 14 12) | 35.85 (49.173) [11.54 to 60.15] | 23.79 (72.638) [-10.59 to 58.17] | 35.86 (47.337) [13.45 to 58.26] | 15.83 (43.151) [-6.54 to 38.20]
  Triglycerides: Change at Week 4 (n=12, 12, 12, 10) | 0.67 (42.470) [-21.35 to 22.68] | 35.67 (80.714) [-6.18 to 77.51] | 24.00 (66.766) [-10.61 to 58.61] | -7.30 (44.144) [-32.89 to 18.29]
  Triglycerides: Change at Week 8 (n= 7, 11, 10, 8) | 48.71 (102.301) [-26.42 to 123.85] | 41.09 (68.405) [3.71 to 78.47] | 12.20 (44.434) [-13.56 to 37.96] | 46.50 (62.198) [4.84 to 88.16]

9. Secondary Outcome: Change From Baseline in Lipid Ratios at Week 2, 4 and 8
Description: The ratio of LDL-C/HDL-C was reported.
Time Frame: Baseline, Week 2, 4, 8 (early termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
ratio
  LDL-C: HDL C; Baseline (n= 14,15,16,14) | 2.35 (0.745) [2.00 to 2.70] | 2.39 (0.915) [1.98 to 2.81] | 2.48 (0.735) [2.16 to 2.80] | 2.37 (0.912) [1.94 to 2.80]
  LDL-C: HDL C; Change at Week 2 (n=13,14,14,12) | 0.02 (0.449) [-0.20 to 0.24] | -0.05 (0.593) [-0.33 to 0.23] | -0.33 (0.384) [-0.51 to -0.14] | -0.03 (0.367) [-0.22 to 0.16]
  LDL C: HDL C; Change at Week 4 (n= 12, 12, 12, 10) | 0.01 (0.218) [-0.10 to 0.12] | 0.11 (0.552) [-0.17 to 0.40] | -0.30 (0.468) [-0.54 to -0.06] | -0.07 (0.813) [-0.54 to 0.40]
  LDL C: HDL C; Change at Week 8 (n=7,11,10, 8) | 0.37 (0.381) [0.09 to 0.65] | 0.32 (0.439) [0.08 to 0.56] | -0.07 (0.324) [-0.26 to 0.12] | -0.04 (0.362) [-0.28 to 0.21]

10. Secondary Outcome: Change From Baseline in High Sensitivity C- Reactive Protein (hsCRP) at Week 1, 2, 3, 4, and 8
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Reference range for measurements is 0-0.5 mg/dL and lower limit of detection is less than (<) 0.015 mg/dL. Any value <0.015 mg/dL is imputed as 0.0075 mg/dL.
Time Frame: Baseline, Week 1, 2, 3, 4, 8 (early termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
mg/dL
  Baseline (n= 14, 15, 16, 14) | 0.6056 (1.05280) [0.1074 to 1.1039] | 0.6718 (0.71527) [0.3465 to 0.9971] | 0.3325 (0.28854) [0.2060 to 0.4589] | 0.4994 (0.43345) [0.2943 to 0.7046]
  Change at Week 1 (n= 14, 15, 16, 14) | -0.1451 (0.37322) [-0.3218 to 0.0315] | -0.5495 (0.66033) [-0.8498 to -0.2492] | -0.2288 (0.26512) [-0.3450 to -0.1127] | -0.3807 (0.49723) [-0.6161 to -0.1454]
  Change at Week 2 (n= 13, 14, 14, 12) | -0.1712 (0.49223) [-0.4145 to 0.0722] | -0.4540 (0.80459) [-0.8349 to -0.0732] | -0.1783 (0.27518) [-0.3085 to -0.0480] | -0.3374 (0.49736) [-0.5952 to -0.0795]
  Change at Week 3 (n= 12, 12, 15, 11) | 0.0323 (0.61746) [-0.2879 to 0.3524] | 1.2447 (5.21627) [-1.4596 to 3.9489] | -0.0471 (0.45332) [-0.2532 to 0.1591] | -0.2214 (0.48102) [-0.4843 to 0.0415]
  Change at Week 4 (n= 11, 12, 12, 10) | -0.0284 (0.64387) [-0.3803 to 0.3235] | -0.4093 (0.83169) [-0.8405 to 0.0218] | 0.1162 (0.95838) [-0.3806 to 0.6131] | -0.0850 (0.63410) [-0.4526 to 0.2826]
  Change at Week 8 (n= 7, 11, 11, 8) | -0.5996 (1.17921) [-1.4656 to 0.2665] | -0.2473 (0.94249) [-0.7623 to 0.2678] | 0.2521 (0.53698) [-0.0413 to 0.5456] | -0.0081 (0.16782) [-0.1205 to 0.1043]

11. Secondary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Epstein-Barr Virus (EBV) Values
Description: EBV samples were collected and changes from baseline were evaluated by the principal investigator (PI) for clinical significance. Clinical significance is levels outside of the normal range (abnormal levels) with clinically apparent viral disease, or that resulted in adverse event (AEs) or required follow-up.
Time Frame: Baseline up to Week 8 (early termination)
Population: The safety analysis population set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Cytomegalovirus (CMV) Values
Description: CMV samples were collected and changes from baseline were evaluated by the PI for clinical significance. Clinical significance is levels outside of the normal range (abnormal levels) with clinically apparent viral disease, or that resulted in AEs or required follow-up.
Time Frame: Baseline up to Week 8 (early termination)
Population: The safety analysis population set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Herpes Simplex Virus Deoxyribonucleic Acid (HSV DNA) Values
Description: HSV DNA samples were collected and changes from baseline were evaluated by the PI for clinical significance. Clinical significance is levels outside of the normal range (abnormal levels) with clinically apparent viral disease, or that resulted in AEs or required follow-up.
Time Frame: Baseline up to Week 8 (early termination)
Population: The safety analysis population set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at Week 1, 2, 3, 4, 5, 6, and 8
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 8 (early termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
millimeter of mercury (mmHg)
  Systolic BP: Baseline (n= 14,15,16,14) | 125.4 (11.77) | 125.5 (11.46) | 124.7 (12.97) | 128.0 (11.50)
  Systolic BP: Change at Week 1 (n= 14, 15, 16, 14) | -2.1 (9.64) | -1.5 (10.94) | 0.6 (8.87) | 2.0 (10.88)
  Systolic BP: Change at Week 2 (n= 13, 13, 14, 10) | -0.3 (6.73) | -1.6 (9.46) | 3.9 (8.01) | -0.4 (7.68)
  Systolic BP: Change at Week 3 (n= 12, 12, 14, 10) | -4.5 (7.09) | -3.3 (7.82) | 6.7 (16.82) | -1.0 (13.65)
  Systolic BP: Change at Week 4 (n= 12, 12, 12, 10) | -2.3 (5.66) | -5.8 (12.40) | 0.2 (7.44) | 1.7 (15.44)
  Systolic BP: Change at Week 5 (n= 11, 12, 12, 9) | -2.9 (9.98) | -0.8 (8.29) | -0.3 (10.37) | 2.0 (18.08)
  Systolic BP: Change at Week 6 (n= 11, 12, 12, 10) | -5.7 (8.95) | -1.3 (7.99) | -2.0 (8.86) | -0.2 (11.37)
  Systolic BP: Change at Week 8 (n= 14, 14, 13, 13) | -2.3 (12.96) | -2.1 (9.61) | -2.1 (7.12) | 3.5 (11.49)
  Diastolic BP: Baseline (n=14,15,16,14) | 77.1 (7.39) | 76.5 (6.84) | 77.4 (9.85) | 79.9 (10.73)
  Diastolic BP: Change at Week 1 (n=14,15,16,14) | 0.0 (6.88) | 0.9 (6.97) | 0.8 (9.99) | 2.0 (10.02)
  Diastolic BP: Change at Week 2 (n=13,13,14,10) | 0.6 (8.08) | 1.5 (8.96) | -0.4 (9.13) | 2.5 (6.08)
  Diastolic BP: Change at Week 3 (n=12,12,14,10) | -0.7 (8.17) | -0.9 (7.50) | 1.1 (7.76) | 0.3 (10.70)
  Diastolic BP Change at Week 4 (n=12,12,12,10) | -2.5 (8.21) | -2.3 (6.61) | 1.2 (5.46) | 2.4 (9.58)
  Diastolic BP: Change at Week 5 (n= 11, 12, 12, 9) | 0.8 (5.13) | 0.0 (5.64) | 0.4 (5.62) | 1.8 (10.32)
  Diastolic BP: Change at Week 6 (n=11,12,12,10) | 0.5 (5.91) | 2.1 (6.36) | -2.8 (5.67) | 0.9 (7.49)
  Diastolic BP: Change at Week 8 (n= 14,14,13,13) | -1.1 (8.12) | -0.6 (6.08) | 1.5 (9.77) | 1.4 (9.26)

15. Secondary Outcome: Change From Baseline in Pulse Rate at Week 1, 2, 3, 4, 5, 6, and 8
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 8 (early termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
beats per minute (bpm)
  Baseline (n= 14, 15, 16, 14) | 67.6 (7.87) | 71.8 (11.85) | 72.2 (11.54) | 72.6 (9.64)
  Change at Week 1 (n= 14, 15, 16, 14) | 1.0 (6.50) | -0.2 (8.51) | 0.0 (10.56) | -4.3 (7.43)
  Change at Week 2 (n= 13, 13, 14, 10) | 2.8 (9.97) | -4.7 (9.39) | -2.4 (8.50) | -2.8 (8.48)
  Change at Week 3 (n= 12, 12, 14, 10) | 4.1 (15.09) | -1.3 (10.76) | -1.5 (11.06) | -2.3 (6.88)
  Change at Week 4 (n= 12, 12, 12, 10) | -1.3 (9.69) | -1.3 (12.89) | -4.7 (10.87) | 0.5 (9.37)
  Change at Week 5 (n= 11, 12, 12, 9) | 5.2 (12.75) | 2.7 (10.44) | -0.8 (10.34) | 7.8 (11.11)
  Change at Week 6 (n= 11, 12, 12, 10) | 4.5 (12.36) | -1.8 (11.46) | 2.4 (8.53) | 4.7 (9.15)
  Change at Week 8 (n= 14, 14, 13, 13) | 0.9 (11.96) | -0.6 (13.87) | -5.3 (11.29) | -1.2 (8.12)

16. Secondary Outcome: Change From Baseline in Respiratory Rate at Week 1, 2, 3, 4, 5, 6, and 8
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 8 (early termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: respiration per minute (resp/min)
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
respiration per minute (resp/min)
  Baseline (n= 14, 15, 16, 13) | 16.2 (1.58) | 17.1 (3.67) | 16.3 (2.44) | 17.0 (2.16)
  Change at Week 1 (n= 14, 15, 16, 13) | -0.5 (1.70) | 0.9 (1.98) | -0.1 (0.81) | -0.3 (1.60)
  Change at Week 2 (n= 13, 13, 14, 9) | -0.5 (1.45) | 0.4 (1.71) | -0.6 (1.82) | 0.7 (2.65)
  Change at Week 3 (n= 12, 12, 14, 9) | -0.3 (0.87) | -0.6 (1.51) | -0.4 (1.69) | 0.2 (1.56)
  Change at Week 4 (n= 12, 12, 12, 9) | 0.2 (2.12) | -0.7 (1.72) | -1.2 (1.75) | 0.0 (1.41)
  Change at Week 5 (n= 11, 12, 12, 8) | 0.1 (1.45) | 0.3 (2.30) | -0.9 (1.78) | -0.6 (1.92)
  Change at Week 6 (n= 11, 12, 12, 9) | -0.4 (0.81) | 0.2 (1.34) | -0.8 (1.54) | -0.2 (1.20)
  Change at Week 8 (n= 14, 14, 13, 12) | -0.3 (1.49) | -0.2 (2.01) | -0.8 (1.30) | -1.0 (1.60)

17. Secondary Outcome: Change From Baseline in Body Temperature at Week 1, 2, 3, 4, 5, 6, and 8
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 8 (early termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
degree celsius
  Baseline (n= 14, 15, 16, 14) | 36.49 (0.363) | 36.59 (0.274) | 36.67 (0.282) | 36.57 (0.433)
  Change at Week 1 (n= 14, 15, 16, 14) | -0.01 (0.264) | -0.03 (0.322) | 0.00 (0.265) | -0.17 (0.271)
  Change at Week 2 (n= 13, 13, 14, 10) | -0.04 (0.366) | -0.22 (0.397) | -0.05 (0.509) | -0.05 (0.273)
  Change at Week 3 (n= 12, 12, 14, 10) | -0.04 (0.391) | -0.21 (0.510) | -0.11 (0.287) | 0.09 (0.501)
  Change at Week 4 (n= 12, 12, 12, 10) | -0.07 (0.467) | -0.21 (0.362) | -0.02 (0.346) | -0.12 (0.477)
  Change at Week 5 (n= 11, 12, 12, 9) | 0.21 (0.316) | 0.07 (0.318) | 0.01 (0.305) | 0.13 (0.443)
  Change at Week 6 (n= 10, 12, 12, 10) | 0.05 (0.328) | -0.00 (0.292) | -0.07 (0.269) | 0.00 (0.390)
  Change at Week 8 (n= 14, 14, 13, 13) | 0.10 (0.332) | -0.01 (0.361) | -0.05 (0.326) | 0.07 (0.426)

18. Secondary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Heart Rate
Time Frame: Baseline up to Week 8 (early termination)
Population: The safety analysis population set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: bpm
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
bpm | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Electrocardiogram (ECG) Parameters
Description: ECG change data was reported as qualitative results, as per change in planned analysis. It was categorized as: normal; abnormal, not clinically significant or abnormal, clinically significant.
Time Frame: Baseline up to Week 8 (early termination)
Population: The safety analysis population set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Number analyzed (Participants) | 14 | 15 | 16 | 14
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-04965842 200 Milligram (mg) Once Daily | PF-04965842 400 mg Once Daily | PF-04965842 200 mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/15 | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 6/14 | 7/15 | 14/16 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | PF-04965842 200 Milligram (mg) Once Daily (N=15) | PF-04965842 400 mg Once Daily (N=16) | PF-04965842 200 mg Twice Daily (N=14)
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | PF-04965842 200 Milligram (mg) Once Daily (N=15) | PF-04965842 400 mg Once Daily (N=16) | PF-04965842 200 mg Twice Daily (N=14)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 5
White blood cell disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 4 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 3
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 5 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to changes in the prioritization of the drug development portfolio and the early termination was not safety related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.